CLINICAL TRIAL: NCT07305740
Title: Online Training After Cancer (On-Trac): Developing An Online Intervention for Cancer Survivors Managing Anxiety
Brief Title: On-Trac: An Online Intervention for Cancer Survivors Managing Anxiety
Acronym: On-Trac
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christopher Recklitis, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-521
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Survivorship; Anxiety
Keywords: Cancer Survivorship; Anxiety
MeSH Terms: conditions — Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: CANCER SURVIVORS AGE 18-39 ON-TRAC SMALL GROUP (Experimental): Participants ages 18-39 will receive a group educational intervention via synchronous video conference that provides strategies for managing anxiety. 1-7 days after attending the educational session, participants will receive a 30- 45 minute individual coaching session by telephone to help them implement strategies to manage anxiety. After the first coaching session each participant will be offered a second (optional) coaching session.
  Interventions: Behavioral: ON-TRAC Education session; Behavioral: ON-TRAC Coaching
- Cohort 2: CANCER SURVIVORS AGE 18-39 ON-TRAC INDIVIDUAL SESSIONS (Experimental): Participants ages 18-39 will receive an individual, 1 on 1, educational intervention via synchronous video conference that provides strategies for managing anxiety. 1-7 days after attending their educational session, participants will receive a 30- 45 minute individual coaching session by telephone to help them implement strategies to manage anxiety. After the first coaching session each participant will be offered a second (optional) coaching session.
  Interventions: Behavioral: ON-TRAC Education session; Behavioral: ON-TRAC Coaching
- Cohort 3: CANCER SURVIVORS AGE 40+ ON-TRAC SMALL GROUP (Experimental): Participants ages 40+ will receive a group educational intervention via synchronous video conference that provides strategies for managing anxiety. 1-7 days after attending the educational session, participants will receive a 30-45 minute individual coaching session by telephone to help them implement strategies to manage anxiety. After the first coaching session each participant will be offered a second (optional) coaching session.
  Interventions: Behavioral: ON-TRAC Education session; Behavioral: ON-TRAC Coaching
- Cohort 4: CANCER SURVIVORS AGE 40+ ON-TRAC INDIVIDUAL SESSIONS (Experimental): Participants ages 18-39 will receive an individual, 1 on 1, educational intervention via synchronous video conference that provides strategies for managing anxiety. 1-7 days after attending their educational session, participants will receive a 30-45 minute individual coaching session by telephone to help them implement strategies to manage anxiety. After the first coaching session each participant will be offered a second (optional) coaching session.
  Interventions: Behavioral: ON-TRAC Education session; Behavioral: ON-TRAC Coaching

INTERVENTIONS:
Behavioral: ON-TRAC Education session — 120 minute educational session on strategies for anxiety delivered via synchronous videoconference session
Behavioral: ON-TRAC Coaching — 30-40 minute individual coaching sessions on implementation of strategies for anxiety

SUMMARY:
This study is evaluating On-Trac (Online Training After Cancer), an online educational intervention to teach adult cancer survivors strategies to address anxiety based on Cognitive-Behavioral Therapy (CBT) and Acceptance Commitment Therapy (ACT)

The name of the study intervention is Online Training After Cancer (On-Trac)

DETAILED DESCRIPTION:
This is a minimal-risk behavioral optimization trial to optimize and refine On-Trac (Online Training After Cancer), an online educational intervention designed to help adult cancer survivors.

The research study procedures include screening for eligibility, questionnaires and interviews.

Participation in the study involves:

* Completing online survey using using a web-based survey platform for baseline assessment
* Taking part in an online, 120 minute, group session via video conference platform and completing an online questionnaire.
* Completing 1-2, 30-40 minute, individual coaching sessions 1-7 days after group educational video session.
* Completing follow-up questionnaire using a web-based survey platform and telephone interview at 4, and 8 weeks after the group education session.
* Participants will receive gift card incentives for completing the brief post-session evaluation and the longer follow-up questionnaires and interview, with a maximum total of $90.

It is expected about 80 people will participate in this research study and will be grouped in four aged based cohorts of 15-20 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* A diagnosis of cancer (except non-melanoma skin cancer) ≥ 12 months prior.
* No active cancer therapy (excluding chemoprevention) in the past 4 months, and no further therapy planned.
* Significant anxiety as evidenced by both of the following

  * Endorsement of the SCID ( Structured Clinical Interview for the DSM-5) Screener Items for Social Anxiety Disorder, Generalized Anxiety Disorder, Agoraphobia, Specific Phobia, or Illness Anxiety Disorder.
  * A score ≥ 6 on the Overall Anxiety Severity and Impairment Scale (OASIS).
* Regular access to the internet.
* Ability to read and write in English.

Exclusion Criteria:

* Significant symptoms of Panic Disorder in the prior 3 months, including anticipatory anxiety of having a future panic attack or avoidance symptoms associated with panic attacks, as assessed by three SCID-5 items from the panic attack disorder module.
* Significant symptoms of Obsessive Compulsive Disorder, as evidenced by any obsessions over the past 3 months, as assessed by three SCID items from the Obsessive Compulsive Disorder module.
* Psychiatric hospitalizations or emergency room visits for psychiatric care in the prior 2 years.
* Any use in the last month of emergent or "rescue" anxiety medication (e.g., Ativan, Xanax, Valium) or self-prescribed substances (i.e., marijuana) at the onset of anxiety symptoms or when entering a situation where they expect to experience anxiety.
* Any significant marijuana use which could impact anxiety symptoms, as evidenced by one of the following:

  * 4 days of marijuana use in any week in the last month
  * 20 milligrams of THC (Tetrahydrocannabinol) products in any week in the last month.
* Participation in any CBT or ACT-based behavioral or education intervention for anxiety in the past 2 years. This includes in-person, asynchronous, and synchronous online anxiety programs, and therapy that includes these skills. This does not include independent use of any self-help materials (i.e., workbooks, books).
* Any impairment (e.g., hearing, visual, cognitive) that interferes with the ability to complete all parts of the study independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in OASIS (Overall Anxiety Severity and Impairment Scale) from baseline to 4 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  OASIS is a 5-item self-report measure, where the total score is obtained as a sum of the individual items. Higher scores are indicative of more severe and impairing anxiety symptoms.
Change in OASIS (Overall Anxiety Severity and Impairment Scale) from baseline to 8 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  OASIS is a 5-item self-report measure, where the total score is obtained as a sum of the individual items. Higher scores are indicative of more severe and impairing anxiety symptoms.
Change in AAQ-2 (Acceptance and Action Questionnaire - Version 2) from baseline to 4 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  AAQ-2 is a 7-item self report measure, where the total score is obtained as a sum of the individual items. Higher scores are indicative of higher psychological inflexibility.
Change in AAQ-2 (Acceptance and Action Questionnaire - Version 2) from baseline to 8 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  AAQ-2 is a 7-item self report measure, where the total score is obtained as a sum of the individual items. Higher scores are indicative of higher psychological inflexibility.
Change in PROMIS-Anxiety from baseline to 4 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  PROMIS-Anxiety is a 7-item self report measure, where the total score is obtained as a sum of the individual items. Higher scores are indicative of greater severity of anxiety symptoms.
Change in PROMIS-Anxiety Short Form 7a (SF-7a) from baseline to 8 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  PROMIS-Anxiety SF-7 is a 7-item self report measure, where the total score is obtained as a sum of the individual items. Higher scores are indicative of greater severity of anxiety symptoms.
Change in IAQ (Illness Anxiety Questionnaire) from baseline to 4 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  IAQ is a 7-item self report measure, with all items adapted from the Short Health Anxiety Inventory (SHAI). The total score is obtained as a sum of the individual items.
Change in IAQ ( Illness Anxiety Questionnaire) from baseline to 8 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  IAQ is a 7-item self report measure, with all items adapted from the Short Health Anxiety Inventory (SHAI). The total score is obtained as a sum of the individual items.
Change in PROMIS-Self Efficacy from baseline to 4 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  SIx PROMIS-Self Efficacy items were selected from the PROMIS item bank for managing chronic conditions - managing emotions. A total score is obtained as a sum of the individual items. Higher scores are indicative of greater self-efficacy for managing emotions.
Change in PROMIS-Self Efficacy from baseline to 8 weeks | Anxiety measures will be collected once at baseline prior to receiving On-Trac intervention, and at follow-up 4 and 8 weeks post-baseline.
  Six PROMIS-Self Efficacy items were selected from the PROMIS item bank for managing chronic conditions - managing emotions. A total score is obtained as a sum of the individual items. Higher scores are indicative of greater self-efficacy for managing emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Recklitis, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: On-Trac Study Coordinator at; ontrac@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu